CLINICAL TRIAL: NCT00676104
Title: Discrete Hypothermia in the Management of Traumatic Brain Injury
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Monique Surles, Designated Investigator, Emory University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 0584-2005
Record Dates: First submitted 2008-05-08; First posted 2008-05-12 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-12

CONDITIONS: Severe Traumatic Brain Injury
Keywords: Traumatic Brain Injury; Trauma; Hypothermia
MeSH Terms: conditions — Brain Injuries, Traumatic; Wounds and Injuries; Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental)
  Interventions: Device: CoolSystems Discrete Cerebral Hypothermia System
- Control (Sham Comparator)
  Interventions: Device: CoolSystems Discrete Cerebral Hypothermia System

INTERVENTIONS:
Device: CoolSystems Discrete Cerebral Hypothermia System — The CoolSystems Discrete Cerebral Hypothermia System (DCHS) will be removed from the patients head after 48 hours.

SUMMARY:
The primary goal of this project is to demonstrate the feasibility and clinical benefits of a new rapid treatment for secondary treatment for secondary brain injury called Discrete Cerebral Hypothermia System by CoolSystems, Inc., Berkley, CA. This device induced hypothermia in the adult brain without significant whole body hypothermia. Discrete Cerebral Hypothermia System holds a great potential for protecting the brain from the devastating secondary complications of trauma without the associated deleterious system effects.

ELIGIBILITY:
Inclusion Criteria:

* Patient is treated for severe traumatic brain injury at Grady Health System, GCS < 8
* Patient is >18 years of age
* Patient requires an Intracranial Pressure (ICP) Probe (part of their routine treatment)
* Patient is able to receive Discrete Cerebral Hypothermia within 48-hours of hospital admission
* Patient and/or guardian must speak English (in order to ensure proper Informed Consent)
* Patient and/or guardian/family must sign an Informed Consent

Exclusion Criteria:

* Unwillingness or inability of patient and/or guardian/ family to sign an informed consent
* Physical placement of cooling cap impedes routine treatment
* Patient has a core body temperature of 36 degrees C or less at time of assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-07; Primary Completion 2007-08 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Perform a comparative analysis of outcome (Glasgow Outcome Score) | Day 1, day 2, day 3, day 7, day 14, day 21, day 28 and 1 month after injury

SECONDARY OUTCOMES:
The effectiveness of the Discrete Cerebral Hypothermia System by CoolSystems in maintaining a significant gradient between the core and brain temperatures in study population. | within 3 days after injury
Functional Independence Measure | Day 1, day 2, day 3, day 7, day 14, day 21, day 28 and 1 month after injury
Mortality | Day 1, day 2, day 3, day 7, day 14, day 21, day 28 and 1 month after injury
Confirm the effectiveness of the Discrete Cerebral System in reducing internal brain temperature | within 3 days after injury

CONTACTS AND LOCATIONS:
Overall Officials: Odette A Harris, MD, MPH, Principal Investigator — Emory University
Locations (1):
- Emory University School of Medicine, Grady Health System campus, Atlanta, Georgia, United States